CLINICAL TRIAL: NCT06963177
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIa Clinical Study to Assess the Efficacy and Safety of GenSci048 in Patients With Moderate to Severe Endometriosis-Associated Pain
Brief Title: A Phase IIa Clinical Study to Assess the Efficacy and Safety of GenSci048 in Patients With Moderate to Severe Endometriosis-Associated Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci048-205
Record Dates: First submitted 2025-04-28; First posted 2025-05-08 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis-related Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GenSci048 (Experimental): GenSci048 subcutaneously (SC) every 4 weeks.
  Interventions: Drug: GenSci048
- Placebo (Placebo Comparator): Administered SC every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GenSci048 — Administered SC.
  Arms: GenSci048
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and efficacy of GenSci048 for moderate to severe endometriosis-associated pain treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal female participants, between 18 and 49 years of age, inclusive, at the time of signing informed consent.
2. Participants must have a diagnosis of endometriosis within 10 years before screening.
3. Have moderate to severe endometrial related pain.
4. Have at least one regular, natural menstrual cycles (ranging from 21 to 35 days (inclusive)) before and during the screening period.
5. Agree to switch from her usual analgesic medication to only that which is permitted in the study from the screening period to the end of treatment and agree to stop using other treatments for endometriosis.
6. Agree to use non-hormonal contraception from the time of signing the informed consent until 4 weeks after the last dose of the study medication.

Exclusion Criteria:

1. Participants who have previously received hysterectomy and/or bilateral oophorectomy, or plan to undergo these procedures during the study period.
2. Participants who suffer from chronic pelvic and/or non-pelvic pain that is not caused by EM and require chronic analgesia or other chronic treatment, which is expected to affect the assessment of EAP.
3. Pelvic ultrasound screening indicating a need for surgery or suspicion of malignancy.
4. Participants with abnormal and undiagnosed vaginal and/or uterine bleeding within 3 months prior to screening.
5. Participants who plan to schedule elective surgery during the study; or those who have had a surgery within 4 months prior to screening and need ongoing pain management.
6. History of severe depression or post-traumatic stress disorder within the two years prior to screening, or history of any other severe mental disorder at any time.
7. History of drug or alcohol abuse within the six months prior to screening.
8. Participants who have participated in any other interventional clinical trial (including clinical trials of drugs and devices) within 1 month prior to screening.
9. Have used a prohibited long-acting anesthetic or immediate-release anesthetic for more than 2 consecutive weeks for the treatment of endometriosis associated pain in the 6 months prior to screening.
10. Participant is pregnant, breast feeding, or planning a pregnancy.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2030-01-06 (Estimated)

PRIMARY OUTCOMES:
Change of dysmenorrhea (DYS) measured by Numeric Rating Scale (NRS) | baseline, week 24
  The NRS for overall endometriosis-associated pain ranges from 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome.
Change of non-menstrual pelvic pain (NMPP) measured by Numeric Rating Scale (NRS) | baseline, week 24
  The NRS for overall endometriosis-associated pain ranges from 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of DYS, NMPP, and dyspareunia (DYSP) measured by Numeric Rating Scale (NRS). The NRS for overall endometriosis-associated pain ranges from 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome. | 52 weeks
Permitted rescue medication use. | 52 weeks
Patient Global Impression of Change, Patient Global Impression of Change (minimum 1, maximum 7, higher score mean a worse outcome). | Week 12、Week 24、Week 52
Adverse Event | up to approximately 56 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China